CLINICAL TRIAL: NCT05319834
Title: Comparative Study Between Vaginal Progesterone Alone or Combined With Aspirin in Prevention of Recurrent Preterm Birth
Acronym: prematurity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Maher, Professor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3/2020/OBG
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: To detect the efficacy and safety of vaginal progesterone alone or combined with aspirin in prevention of recurrent PTB.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants and investigators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progesterone with asprin (Active Comparator): The included women will be randomly allocated to prophylactically receive either vaginal progesterone at a dose of 200 mg (prontogest 200mg every 12 hr) combined with oral aspirin at a dose of 100mg once daily both at the same time (group1),
  Interventions: Drug: Aspirin tablet
- Progesterone and placebo (Placebo Comparator): vaginal progesterone (prontogest 200mg every 12 hr) and oral placebo (manufactured in a standard way to have the same size and shape of asprin tablet) also at the same time (group 2).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin tablet — group1: oral aspirin at a dose of 100mg once daily at the same time with progesterone
  Other Names: group 1 intervention
  Arms: Progesterone with asprin
Drug: Placebo — group 2: oral placebo once daily at the same time with progesterone
  Other Names: group 2 intervention
  Arms: Progesterone and placebo

SUMMARY:
This is a double blinded randomized placebo controlled clinical trial to detect the efficacy and safety of vaginal progesterone alone or combined with aspirin in prevention of recurrent PTB.

DETAILED DESCRIPTION:
The included women will be randomly allocated to prophylactically receive either vaginal progesterone at a dose of 200 mg (prontogest 200mg every 12 hr) combined with oral aspirin at a dose of 100mg once daily both at the same time (group1), or vaginal progesterone (prontogest 200mg every 12 hr) and oral placebo (manufactured in a standard way to have the same size and shape of asprin tablet) also at the same time (group 2).

ELIGIBILITY:
Inclusion Criteria:

1. Women of any age
2. Any parity
3. Healthy singleton pregnancy
4. History suggestive of one or more previous PTB
5. Current pregnancy (16-20) weeks gestation.

Exclusion Criteria:

1. Multifetal pregnancy.
2. History of ante partum PROM.
3. Cervical Incompetence or current cervical cerclage.
4. Known fetal anomaly.
5. Hypertension requiring medications.
6. History of Thrombo-embolic disorders.
7. Known allergy to progesterone or asprin.
8. Known liver disease.
9. Established preterm labor
10. Short cervix

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who will deliver before 34 weeks gestation. | 18 month
  Number of participants who have preterm delivery before 34 weeks gestation

SECONDARY OUTCOMES:
The number of participants who have prolongation of pregnancy after 34 till 37 weeks gestation | 18 months
  Number of participants who will deliver after 34w gestation and neonatal outcomes
Neonatal outcomes | 18 months
  Neonatal birth weight Admission to NICU Neonatal complications

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No